CLINICAL TRIAL: NCT02553200
Title: Study of Breathing Exercise With Oscillated Inspiratory Loading (OIS) and Oscillated Positive Expiratory Pressure (OPEP) for Airway Secretion Clearance and Lung Function in Intubated Patients, Both With and Without Mechanical Ventilatory Support
Brief Title: The Efficacy of Breathing Exercise With BreatheMAX Device on Airway Secretion Clearance and Lung Function
Acronym: BMACPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sujittra Kluayhomthong, 123 Moo 16 Mittapap Road Nai-Muang, Muang District Khon Kaen 40002, Thailand, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KKU
Record Dates: First submitted 2015-05-13; First posted 2015-09-17 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2015-12

CONDITIONS: Bronchial Secretion Retention
Keywords: intubated patients; secretion clearance; lung function; breathing exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BreatheMAX (OPEP) (Active Comparator): for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Interventions: Device: BreatheMAX (OPEP)
- BreatheMAX (OIS and OPEP) (Experimental): for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Interventions: Device: BreatheMAX (OIS and OPEP)
- BreatheMAX (unload and non-oscillated) (Sham Comparator): inspiratory and expiratory breathing exercise for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Interventions: Device: BreatheMAX (unload and non-oscillated)

INTERVENTIONS:
Device: BreatheMAX (OPEP) — for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Arms: BreatheMAX (OPEP)
Device: BreatheMAX (OIS and OPEP) — for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Arms: BreatheMAX (OIS and OPEP)
Device: BreatheMAX (unload and non-oscillated) — for 10 breathes/set, 10 sets/day and rest 1 minute between set
  Arms: BreatheMAX (unload and non-oscillated)

SUMMARY:
The efficacy of breathing exercise with oscillated inspiratory loading and oscillated positive expiratory pressure for airway secretion clearance and lung function in intubated patients, both with and without mechanical ventilation dependence

DETAILED DESCRIPTION:
Effective strategies to increase mucus clearance rate has been suggested to depend on 4 factors.

1. Oscillation at proper frequency.
2. Lung volume and airway opening.
3. Expiratory flow rate or expiratory bias.
4. Humidifying of inspired air.

Multifunctional breathing device, the BreatheMAX, is the only breathing device made in Thailand. The BreatheMAX device possess many properties or techniques that benefit for respiratory care particularly 3 in 4 mechanisms for secretion clearance. The unique important aspect is the simultaneously providing several beneficial effects in one breath which are 1) Oscillation in the range of ciliary beat frequency 2) Biofeedback of respiratory effort that could encourage the deeper breathing performance, 3) Humidifier of inspired air, 4) Loaded breathing for inspiratory muscle training and generate PEP. These 4 functions would be very useful for increase secretion clearance particularly in more peripheral airway which are the most difficult to be cleared and be a risk of atelectasis and infection in patients with MV whose natural secretion clearance mechanisms are compromised, respiratory muscle weakness weak and low immunity.

Therefore, the combination of inspiratory and expiratory breathing exercise through the BreatheMAX breathing device may increase or promote more secretion clearance and improve lung function than expiratory breathing exercise alone in intubated patients, both with and without mechanical ventilation dependence

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients (with and without mechanical ventilator support) with secretion 1.5 ml/h, If the patients are breathing with mechanical ventilation, the PEEP level must be less than 6 centimeter of water and one of following
* Clinical and radiologic diagnosis of pulmonary infection
* Acute or chronic airway inflammation disease such as pneumonia, bronchiectasis, chronic obstructive pulmonary disease or chronic bronchitis and at least one sign of secretion accumulation in bronchial such as medium-coarse crackle, wheezing, persistent rhonchi and decrease breath sound
* Stable of cardiopulmonary function at least 2 days before the study and the patients don't receive the vasopressors drug within 5 days before collects the data
* Stable of hydration status or positive fluid balance at least 2 days before collects the data
* Ability to breathe or tolerate spontaneously breathing trial with T-piece at least 2 minutes with fraction of inspired oxygen less than 0.4 and without developing hypoxemia
* Good conscious and well cooperation

Exclusion Criteria:

* Pneumothorax (nontreated)
* Massive hemoptysis
* Acute myocardial infarction (with angina chest pain)
* High intracranial pressure (>20 mm Hg)
* Major arrhythmia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
change from baseline in secretion wet weight (gram) between 3 hours before and after breathing exercise program | the secretion will be collected between 3 hours before start breathing exercise program and 3 hours after end of breathing exercise program in each day
  The mucus secretion will be collected by nursing staff using sterile suctioning technique via tracheostomy (TT) or endotracheal (ET) tube, without adding any saline or sterile water, the timing of suction procedure depend on the secretion sound in the ET and TT tube.

SECONDARY OUTCOMES:
change from baseline in dynamic compliance (Cdyn) at end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP, VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * the data will be recorded from the mechanical ventilator monitoring during the patients breathing with mechanical ventilation (MV) at least 1 minute
change from baseline in peak inspiratory pressure (PIP) at end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP,VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * the data will be recorded from the mechanical ventilator monitoring during the patients breathing with mechanical ventilation at least 1 minute
change from baseline in expired minute ventilation (VE) at end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP, VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * the wright respirometer will be connected with ET or TT tube during spontaneous breathing (off MV) for 1 minute, three measurement will be measured and rest 1 minute by using mechanical ventilation
change from baseline in slow vital capacity (SVC) at end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP, VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * the wright respirometer will be connected with ET or TT tube during spontaneous breathing (off MV), three measurement will be measured and rest 1 minute by using mechanical ventilation
change from baseline in lung sound at the end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP, PNIP, VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * the electronic stethoscope will be used to record the lung sound in each area during breathing with mechanical ventilation
change from baseline in Rating of Perceived Exertion (RPE) and Rating of Perceived Breathlessness (RPB) at the end of breathing exercise program | within 30 minutes before breathing exercise and 30 minute after breathing exercise
  * as follows: Cdy, PIP, VE, SVC, PEFR, Lung sound, RPE and RPB and cardiopulmonary response
  * using the dyspnea and exertion scale
change from baseline in heart rate at the end of breathing exercise program | 5 minutes before breathing exercise and during breathing exercise and 5 minute after breathing exercise
  the data will be recorded every minute
change from baseline in partial pressure of oxygen saturation at the end of breathing exercise program | 5 minutes before breathing exercise and during breathing exercise and 5 minute after breathing exercise
  the data will be recorded every minute
change from baseline in respiratory rate at the end of breathing exercise program | 5 minutes before breathing exercise and during breathing exercise and 5 minute after breathing exercise
  the data will be recorded every minute
change from baseline in blood pressure at the end of breathing exercise program | 5 minutes before breathing exercise and 5 minute after breathing exercise

CONTACTS AND LOCATIONS:
Overall Officials: Chulee Jones, PhD, Principal Investigator — The Faculty of Associated Medical Sciences Khon Kaen University 123 Moo 16 Mittapap Road Nai-Muang, Muang District Khon Kaen 40002, Thailand
Locations (1):
- Sujittra Kluayhomthong, Khon Kaen, Thailand